CLINICAL TRIAL: NCT07125833
Title: A Randomized Pilot Trial for Cryoneurolysis of the Suprascapular Nerve for Perioperative Pain Control After Receiving a Reverse Total Shoulder Arthroplasty
Brief Title: Cryoneurolysis of the Suprascapular Nerve for Perioperative Pain Control After Receiving a Reverse Total Shoulder Arthroplasty (RTSA)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: North Texas Medical Research Institute, PLLC (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT 24-376
Record Dates: First submitted 2025-08-01; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Degenerative Joint Disease of Shoulder
Keywords: cryoneurolysis; degenerative joint disease; reverse shoulder arthroplasty
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Intervention Model Description: Randomization The design of this trial will utilize a 1:1 randomization schema. Randomization will be performed by an online randomization tool from the National Cancer Institute (https://ctrandomization.cancer.gov/home/). This randomization list will be kept with the study trial documents in a secured location and initially blinded from the primary research team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control (Active Comparator): Those that do not receive cryoneurolysis of the suprascapular nerve prior to RTSA
  Interventions: Other: No cryoneurolysis
- Intervention (Experimental): Those that do receive cryoneurolysis of the suprascapular nerve prior to RTSA
  Interventions: Device: Cryoneurolysis

INTERVENTIONS:
Device: Cryoneurolysis — Cryoneurolysis of the suprascapular nerve
  Arms: Intervention
Other: No cryoneurolysis — Control Group
  Arms: Control

SUMMARY:
The main purpose of this research is to find out if a treatment called cryoneurolysis can reduce pain after reverse total shoulder replacement surgery. This treatment uses cold to temporarily block a nerve in the shoulder. The study will compare people who receive the treatment to those who do not, to see if it helps lower pain and reduce the need for opioid pain medications after a reverse total shoulder surgery (RTSA).

DETAILED DESCRIPTION:
Randomized controlled, pilot clinical trial to assess the administration of and feasibility for cyroneurolysis of the suprascapular nerve in the pre-operative setting for patients that will receive a reverse total shoulder arthroplasty (RTSA). Our primary research hypothesis is that patients who receive the intervention treatment of cryoneurolysis will experience decreased opioid usage compared to the control patient population. Primary: Assess the effectiveness and feasibility of cryoneurolysis of the suprascapular nerve performed pre-operatively for RTSA patients in reduction of the cumulative opioid consumption in the post-operative of 90 days as measured by morphine milligram equivalents (MMEs) compared to those patients who did not receive the intervention prior to a RTSA.

Secondary: Assess the effectiveness of cryoneurolysis of the suprascapular nerve performed pre-operatively for RTSA patients to show:

1. a decreased pain score as measured by a Pain Assessment Documentation Tool (PADT) score
2. increased range of motion
3. increased patient reported outcome scores via the American Shoulder and Elbow Surgeons (ASES) shoulder score when compared to those that did not receive any intervention prior to a RTSA?

ELIGIBILITY:
Inclusion Criteria:

* Male patients or female who are not pregnant and do not plan on future pregnancy during trial participation
* between 30-85 years of age
* BMI less than or equal to 45
* Currently setup for an elective primary reverse total shoulder arthroplasty due to primary osteoarthritis
* Ability to provide informed consent to participate in the clinical trial
* Ability to understand and communicate in English
* Willingness to comply with all study procedures

Exclusion Criteria:

* poorly controlled comorbidities that would not allow surgical intervention such as poorly controlled diabetes (HbA1C > 8.0) renal insufficiency (eGFR <60) poorly controlled CV disease such as CHF that is NYHA class 3 and 4
* inability to receive the intervention including contraindications:
* Cryoglobulinemia, paroxysmal cold hemoglobinuria, cold urticaria, Raynaud's disease, and open and/or infected wounds at or near the treatment site
* patients with history of total joint infection ever or any infection in the last 6 months
* ASA score >3 and Outpatient Arthroplasty Risk Assessment (OARA; medical risk stratification scoring system to help determine day surgery vs inpatient)1 score > 80.
* previous cryoneurolysis of the suprascapular nerve-utilization of supplemental/holistic methods specifically for pain control (e.g. cannabidiol). This will be discontinued 30 days prior to RTSA and will not be used during the duration of study participation. This will be evaluated by the Principal Investigator and study team prior to consent.
* significant anti-coagulation usage (other than aspirin) 7 days prior to treatment
* CV surgery within the last 6 months
* significant neurologic compromise (acquired or congenital/genetic) of the upper extremity to be operated on or underlying neurologic condition that would confound results in the opinion of the investigator such as a

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint for the primary objective would be decreased opioid utilization in the post-operative period after a reverse total shoulder arthroplasty (RTSA) as measured by Morphine Milligram Equivalents (MME). | 90 days
  Pain medication usage as recorded by MME. MME is calculated by multiplying the opioid dose (in mg) by a drug-specific conversion factor (e.g., oxycodone × 1.5, hydromorphone × 4, fentanyl patch mcg/hr × 2.4).
  In research and clinical practice, MME helps quantify total opioid burden, assess risk for overdose, and standardize analgesic reporting in clinical trials. Higher daily MMEs are associated with increased adverse event risk. This will be recorded at every clinical visit.

SECONDARY OUTCOMES:
Decreased Pain Assessment and Documentation Tool (PADT) scores | 90 days
  The Pain Assessment and Documentation Tool (PADT) is a clinician-administered instrument for consistent evaluation of chronic pain in patients on analgesic therapy. It assesses: Pain Intensity (0-10 Numeric Rating Scale: 0 = no pain, 10 = worst pain imaginable; patient rates worst, least, average, and current pain over a set period), Impact on Function (interference with activity, mood, work, relationships, sleep, enjoyment of life, rated 0-10), Adverse Effects/Risk (presence and severity of medication side effects, aberrant behaviors), and Therapeutic Response (clinician summary of effectiveness and regimen changes). In clinical trials, the PADT is used at baseline and follow-up to capture pain severity, functional outcomes, and tolerability, ensuring standardized, reproducible data for efficacy and safety evaluation and is completed by the clinician and participant.
Improved range of motion (ROM) of the shoulder as measured by the investigators and physical therapy documentation | 90 days
  Improved ROM as measured by the investigators and physical therapy documentation. This will be tracked for every therapy and clinical visit. The goal is improved ROM as the patient progresses in the acute phase of post-surgical care.
Decreased American Shoulder and Elbow Surgeons (ASES) patient reported outcomes | 90 days
  The American Shoulder and Elbow Surgeons (ASES) Standardized Shoulder Assessment Form is a validated tool combining patient-reported and clinician-assessed measures to evaluate shoulder function. The patient-reported section (50 points) assesses pain using a 0-10 Visual Analog Scale (converted to 50 points) and function via 10 daily activity questions (scored 0 = unable to do, 3 = no difficulty; summed and scaled to 50 points). The clinician-assessed section includes range of motion and physical exam findings but is not used in the primary score calculation. The total ASES score (0-100) is the sum of pain and function subscores, with higher scores indicating better shoulder function. In clinical trials, the ASES is administered at baseline and follow-up to quantify changes in pain and functional capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad U Burney, MD, Principal Investigator — North Texas Medical Research Institute, PLLC
Locations (1):
- Orthopaedic Specialists of Dallas, Rockwall, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Proprietary

REFERENCES:
- [Background] MacRae F, Boissonnault E, Hashemi M, Winston P. Bilateral Suprascapular Nerve Cryoneurolysis for Pain Associated With Glenohumeral Osteoarthritis: A Case Report. Arch Rehabil Res Clin Transl. 2023 Jan 25;5(1):100256. doi: 10.1016/j.arrct.2023.100256. eCollection 2023 Mar. PMID 36968166
- [Background] Best MJ, Aziz KT, Wilckens JH, McFarland EG, Srikumaran U. Increasing incidence of primary reverse and anatomic total shoulder arthroplasty in the United States. J Shoulder Elbow Surg. 2021 May;30(5):1159-1166. doi: 10.1016/j.jse.2020.08.010. Epub 2020 Aug 26. PMID 32858194
- [Background] Trescot AM. Cryoanalgesia in interventional pain management. Pain Physician. 2003 Jul;6(3):345-60. PMID 16880882